CLINICAL TRIAL: NCT00614380
Title: An Open Label Follow-up Trial of the Efficacy and Safety of Chronic Administration of the Combination of Telmisartan 40mg + Amlodipine 5mg or the Combination of Telmisartan 80mg + Amlodipine 5mg Tablets Alone or in Combination With Other Antihypertensive Medications in Patients With Hypertension.
Brief Title: Open Label Study Telmisartan and Amlodipine in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 1235.7; EUDRACT2007-002410-19
Record Dates: First submitted 2008-01-28; First posted 2008-02-13 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine

INTERVENTIONS:
Drug: telmisartan/amlodipine 40/5 mg fixed combination
Drug: telmisartan/amlodipine 80/5 mg fixed combination

SUMMARY:
The primary objective of this trial is to assess the efficacy and safety of the fixed dose combinations telmisartan 40 mg / amlodipine 5 mg (T40/A5) or telmisartan 80 mg / amlodipine 5 mg (T80/A5) during long-term open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged at least 18 years
2. diagnosis of essential hypertension and blood pressure not adequately controlled before enrolment in the preceding trial.
3. failure to respond to six weeks treatment with Amlodipine 5 mg in the run-in period of the preceding trial.

Exclusion Criteria:

1. pre-menopausal women who are not surgically sterile; or are nursing or pregnant; or are not practising acceptable means of birth control or do not plan to continue using acceptable means of birth control throughout the study
2. development of any medical condition in the preceding trial that in the investigator's opinion could be worsened by treatment with either Telmisartan 40 mg/Amlodipine 5 mg or Telmisartan 80 mg/Amlodipine 5 mg
3. discontinuation from the preceding trial because of any adverse event or any other reason
4. known or suspected secondary hypertension
5. mean seated Systolic Blood Pressure => 180 mmHg and/or mean seated Diastolic Blood Pressure => 120 mmHg at any visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (122):
- Belgium (7):
  - 1235.7.32004 Boehringer Ingelheim Investigational Site, Aywaille
  - 1235.7.32010 Boehringer Ingelheim Investigational Site, Gozée
  - 1235.7.32008 Boehringer Ingelheim Investigational Site, Linkebeek
  - 1235.7.32003 Boehringer Ingelheim Investigational Site, Mol
  - 1235.7.32007 Boehringer Ingelheim Investigational Site, Natoye
  - 1235.7.32002 Boehringer Ingelheim Investigational Site, Tienen
  - 1235.7.32005 Boehringer Ingelheim Investigational Site, Turnhout
- Canada (12):
  - 1235.7.20001 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 1235.7.20011 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1235.7.20007 Boehringer Ingelheim Investigational Site, Bay Roberts, Newfoundland and Labrador
  - 1235.7.20005 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 1235.7.20008 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1235.7.20013 Boehringer Ingelheim Investigational Site, Corunna, Ontario
  - 1235.7.20014 Boehringer Ingelheim Investigational Site, Etobicoke, Ontario
  - 1235.7.20010 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1235.7.20012 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1235.7.20009 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1235.7.20006 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1235.7.20003 Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
- Denmark (8):
  - 1235.7.45002 Boehringer Ingelheim Investigational Site, Birkerød
  - 1235.7.45005 Boehringer Ingelheim Investigational Site, Haderslev
  - 1235.7.45008 Boehringer Ingelheim Investigational Site, Herning
  - 1235.7.45009 Boehringer Ingelheim Investigational Site, Hinnerup
  - 1235.7.45001 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 1235.7.45006 Boehringer Ingelheim Investigational Site, Rødovre Municipality
  - 1235.7.45003 Boehringer Ingelheim Investigational Site, Vaerløse
  - 1235.7.45007 Boehringer Ingelheim Investigational Site, Vildbjerg
- Finland (4):
  - 1235.7.35003 Boehringer Ingelheim Investigational Site, Joensuu
  - 1235.7.35004 Boehringer Ingelheim Investigational Site, Joensuu
  - 1235.7.35001 Boehringer Ingelheim Investigational Site, Turku
  - 1235.7.35002 Boehringer Ingelheim Investigational Site, Turku
- France (44):
  - 1235.7.3301H Boehringer Ingelheim Investigational Site, Aigrefeuille S/Maine
  - 1235.7.3306C Boehringer Ingelheim Investigational Site, Angers
  - 1235.7.3309B Boehringer Ingelheim Investigational Site, Angers
  - 1235.7.3309C Boehringer Ingelheim Investigational Site, Angers
  - 1235.7.3309E Boehringer Ingelheim Investigational Site, Angers
  - 1235.7.3309D Boehringer Ingelheim Investigational Site, Avrillé
  - 1235.7.3309A Boehringer Ingelheim Investigational Site, Beaucouzé
  - 1235.7.3305A Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 1235.7.3306D Boehringer Ingelheim Investigational Site, Briollay
  - 1235.7.3308B Boehringer Ingelheim Investigational Site, Cholet
  - 1235.7.3308F Boehringer Ingelheim Investigational Site, Cholet
  - 1235.7.3302C Boehringer Ingelheim Investigational Site, Garchizy
  - 1235.7.3303C Boehringer Ingelheim Investigational Site, Grandchamps
  - 1235.7.3302D Boehringer Ingelheim Investigational Site, Guérigny
  - 1235.7.3310A Boehringer Ingelheim Investigational Site, Jarny
  - 1235.7.3301L Boehringer Ingelheim Investigational Site, La Chapelle /s Erdre
  - 1235.7.3301J Boehringer Ingelheim Investigational Site, La Chapelle-sur-Erdre
  - 1235.7.3304A Boehringer Ingelheim Investigational Site, La Fresnais
  - 1235.7.3308E Boehringer Ingelheim Investigational Site, La Jubaudière
  - 1235.7.3301G Boehringer Ingelheim Investigational Site, La Montagne
  - 1235.7.3307D Boehringer Ingelheim Investigational Site, Le Mesnil-en-Vallée
  - 1235.7.3301E Boehringer Ingelheim Investigational Site, Le Temple-de-Bretagne
  - 1235.7.3309F Boehringer Ingelheim Investigational Site, Les Ponts-de-Cé
  - 1235.7.3305B Boehringer Ingelheim Investigational Site, Louvigné Le Bais
  - 1235.7.3307E Boehringer Ingelheim Investigational Site, Mouliherne
  - 1235.7.3306A Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 1235.7.3307A Boehringer Ingelheim Investigational Site, Mûrs-Erigné
  - 1235.7.3301A Boehringer Ingelheim Investigational Site, Nantes
  - 1235.7.3301B Boehringer Ingelheim Investigational Site, Nantes
  - 1235.7.3301D Boehringer Ingelheim Investigational Site, Nantes
  - 1235.7.3301M Boehringer Ingelheim Investigational Site, Nantes
  - 1235.7.3302A Boehringer Ingelheim Investigational Site, Nevers
  - 1235.7.3302F Boehringer Ingelheim Investigational Site, Nevers
  - 1235.7.3301I Boehringer Ingelheim Investigational Site, Nort-sur-Erdre
  - 1235.7.3301C Boehringer Ingelheim Investigational Site, Orvault
  - 1235.7.3307F Boehringer Ingelheim Investigational Site, Parçay-les-Pins
  - 1235.7.3301F Boehringer Ingelheim Investigational Site, Saint Aubin Les Châteaux
  - 1235.7.3306F Boehringer Ingelheim Investigational Site, Saint-Georges-de-Montaigu
  - 1235.7.3304B Boehringer Ingelheim Investigational Site, Saint-Ouen-la-Rouërie
  - 1235.7.3301N Boehringer Ingelheim Investigational Site, Sautron
  - 1235.7.3306B Boehringer Ingelheim Investigational Site, Segré
  - 1235.7.3306E Boehringer Ingelheim Investigational Site, Thouars
  - 1235.7.3304C Boehringer Ingelheim Investigational Site, Tinténiac
  - 1235.7.3308A Boehringer Ingelheim Investigational Site, Vihiers
- Netherlands (8):
  - 1235.7.31008 Boehringer Ingelheim Investigational Site, Beerzerveld
  - 1235.7.31006 Boehringer Ingelheim Investigational Site, Bennebroek
  - 1235.7.31004 Boehringer Ingelheim Investigational Site, Hoogwoud
  - 1235.7.31003 Boehringer Ingelheim Investigational Site, Musselkanaal
  - 1235.7.31007 Boehringer Ingelheim Investigational Site, Nijverdal
  - 1235.7.31001 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1235.7.31005 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 1235.7.31010 Boehringer Ingelheim Investigational Site, Voerendaal
- Norway (4):
  - 1235.7.47001 Boehringer Ingelheim Investigational Site, Ålesund
  - 1235.7.47002 Boehringer Ingelheim Investigational Site, Bergen
  - 1235.7.47003 Boehringer Ingelheim Investigational Site, Hamar
  - 1235.7.47004 Boehringer Ingelheim Investigational Site, Oslo
- Philippines (8):
  - 1235.7.63006 Boehringer Ingelheim Investigational Site, Makati City
  - 1235.7.63001 Boehringer Ingelheim Investigational Site, Manila
  - 1235.7.63002 Boehringer Ingelheim Investigational Site, Manila
  - 1235.7.63009 Boehringer Ingelheim Investigational Site, Manila
  - 1235.7.63008 Boehringer Ingelheim Investigational Site, Pasay
  - 1235.7.63005 Boehringer Ingelheim Investigational Site, Pasig
  - 1235.7.63003 Boehringer Ingelheim Investigational Site, Quezon City
  - 1235.7.63007 Boehringer Ingelheim Investigational Site, Quezon City
- South Africa (10):
  - 1235.7.27003 Boehringer Ingelheim Investigational Site, Boksburg
  - 1235.7.27006 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.7.27009 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.7.27010 Boehringer Ingelheim Investigational Site, Cape Town
  - 1235.7.27004 Boehringer Ingelheim Investigational Site, Durban
  - 1235.7.27007 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1235.7.27008 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1235.7.27001 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1235.7.27005 Boehringer Ingelheim Investigational Site, Lenasia
  - 1235.7.27002 Boehringer Ingelheim Investigational Site, Pretoria
- South Korea (8):
  - 1235.7.82007 Boehringer Ingelheim Investigational Site, Busan
  - 1235.7.82001 Boehringer Ingelheim Investigational Site, Daegu
  - 1235.7.82006 Boehringer Ingelheim Investigational Site, Daejeon
  - 1235.7.82004 Boehringer Ingelheim Investigational Site, Gangwon-Do
  - 1235.7.82008 Boehringer Ingelheim Investigational Site, Gwangju
  - 1235.7.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.7.82003 Boehringer Ingelheim Investigational Site, Seoul
  - 1235.7.82005 Boehringer Ingelheim Investigational Site, Seoul
- Sweden (5):
  - 1235.7.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1235.7.46003 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1235.7.46005 Boehringer Ingelheim Investigational Site, Luleå
  - 1235.7.46004 Boehringer Ingelheim Investigational Site, Rättvik
  - 1235.7.46001 Boehringer Ingelheim Investigational Site, Stockholm
- Taiwan (4):
  - 1235.7.88605 Boehringer Ingelheim Investigational Site, Changhua
  - 1235.7.88608 Boehringer Ingelheim Investigational Site, Hualien City
  - 1235.7.88601 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1235.7.88603 Boehringer Ingelheim Investigational Site, Taichung

REFERENCES:
- [Derived] Neldam S, Edwards C, Lang M, Jones R; TEAMSTA-5 and TEAMSTA-10 Investigators. Long-Term Tolerability and Efficacy of Single-Pill Combinations of Telmisartan 40-80 mg Plus Amlodipine 5 or 10 mg in Patients Whose Blood Pressure Was Not Initially Controlled by Amlodipine 5-10 mg: Open-Label, Long-Term Follow-Ups of the TEAMSTA-5 and TEAMSTA-10 Studies. Curr Ther Res Clin Exp. 2012 Feb;73(1-2):65-84. doi: 10.1016/j.curtheres.2012.02.004. PMID 24653513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Started | 564 | 206 | 25 | 181
Completed | 529 | 198 | 24 | 179
Not Completed | 35 | 8 | 1 | 2
Not completed — Adverse Event | 14 | 4 | 0 | 0
Not completed — Lost to Follow-up | 6 | 1 | 0 | 0
Not completed — Non compliant with the protocol | 12 | 2 | 1 | 2
Not completed — Consent withdrawn | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive | Total
Number analyzed (Participants) | 564 | 206 | 25 | 181 | 976
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (10.9) | 52.9 (10.6) | 54.4 (10.8) | 52.4 (9.6) | 53.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 72 | 8 | 45 | 365
  Male | 324 | 134 | 17 | 136 | 611

OUTCOME MEASURES:

1. Primary Outcome: Trough Seated Diastolic Blood Pressure (DBP) Control
Description: The number of patients who reach the target DBP of <90mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: The full analysis set of patients. All patients who took at least one dose of study medication and have at least one on treatment BP measurement 20-30 hours post dose
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 553 | 206 | 25 | 181
Participants
  Yes (DBP<90 mmHg) | 504 | 160 | 19 | 84
  No (DBP>=90 mmHg) | 49 | 46 | 6 | 97
Statistical Analysis 1: Comparison: Telmisartan 40mg and Amlodipine 5mg vs Telmisartan 80mg and Amlodipine 5mg; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.34, 95% CI [0.22 to 0.53]
Statistical Analysis 2: Comparison: Telmisartan 40mg and Amlodipine 5mg vs Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.31, 95% CI [0.12 to 0.81]
Statistical Analysis 3: Comparison: Telmisartan 40mg and Amlodipine 5mg vs Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.08, 95% CI [0.06 to 0.13]
Statistical Analysis 4: Comparison: Telmisartan 80mg and Amlodipine 5mg vs Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.91, 95% CI [0.34 to 2.41]
Statistical Analysis 5: Comparison: Telmisartan 80mg and Amlodipine 5mg vs Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.25, 95% CI [0.16 to 0.39]
Statistical Analysis 6: Comparison: Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive vs Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.27, 95% CI [0.10 to 0.72]

2. Secondary Outcome: Trough Seated Systolic Blood Pressure (SBP) Control
Description: The number of patients who reach the target SBP of <140mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 553 | 206 | 25 | 181
Participants
  Yes (SBP<140 mmHg) | 440 | 142 | 16 | 89
  No (SBP>=140 mmHg) | 113 | 64 | 9 | 92

3. Secondary Outcome: Change From Baseline in Trough Seated Diastolic Blood Pressure
Description: Change from baseline to the end of study in trough DBP. Baseline is defined as visit 3 of trial 1235.5.
Time Frame: End of study (34 weeks or last value on treatment)
Population: All patients who took at least one dose of study medication, have a trough baseline measurement (Visit 3 1235.5) and at least one on treatment BP measurement 20-30 hours post dose
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 549 | 203 | 24 | 176
mmHg | -14.18 (0.31) | -12.64 (0.52) | -9.47 (1.51) | -10.17 (0.56)

4. Secondary Outcome: Change in DBP From Last Available Trough in 1235.5 to Last Available Trough in 1235.7
Description: The difference between the last available troughs represents the additional reduction in DBP in this study
Time Frame: End of study (34 weeks or last value on treatment)
Population: Full Analysis Set (FAS) included patients who took at least one dose of study medication and have at least one on treatment BP measurement
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 545 | 203 | 24 | 180
mmHg | -3.54 (0.33) | -5.52 (0.55) | -5.51 (1.59) | -5.74 (0.58)

5. Secondary Outcome: Change From Baseline in Trough Seated Systolic Blood Pressure
Description: Change from baseline to the end of study in trough SBP. Baseline is defined as visit 3 of trial 1235.5.
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 549 | 203 | 24 | 176
mmHg | -17.79 (0.52) | -15.91 (0.86) | -12.6 (2.5) | -14.04 (0.92)

6. Secondary Outcome: Change in SBP From Last Available Trough in 1235.5 to Last Available Trough in 1235.7
Description: The difference between the last available troughs represents the additional reduction in SBP in this study
Time Frame: End of study (34 weeks or last value on treatment)
Population: All patients who took at least one dose of study medication, have a trough baseline measurement (Last value on treatment in 1235.5) and at least one on treatment BP measurement 20-30 hours post dose
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 545 | 203 | 24 | 180
mmHg | -4.14 (0.5) | -5.62 (0.83) | -3.6 (2.41) | -7.17 (0.88)

7. Secondary Outcome: Trough Seated DBP Response
Description: The number of patients who reach the target DBP of <90mmHg or had a reduction in DBP >= 10mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 553 | 206 | 25 | 181
Participants
  Yes (Responder) | 504 | 171 | 19 | 108
  No (Non-responder) | 45 | 32 | 5 | 68

8. Secondary Outcome: Trough Seated SBP Response
Description: The number of patients who reach the target SBP of <140mmHg or had a reduction in SBP >= 15 mmHg
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 553 | 206 | 25 | 181
Participants
  Yes (Responder) | 490 | 179 | 18 | 128
  No (Non-responder) | 59 | 24 | 6 | 48

9. Secondary Outcome: Trough Blood Pressure (BP) Normality Classes
Description: The number of patients who reach predefined BP categories
Time Frame: End of study (34 weeks or last value on treatment)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg | Telmisartan 40mg and Amlodipine 5mg + add-on Antihypertensive | Telmisartan 80mg and Amlodipine 5mg + add-on Antihypertensive
Number analyzed (Participants) | 553 | 206 | 25 | 181
Participants
  Optimal (SBP<120 and DBP<80 mmHg) | 67 | 4 | 1 | 6
  Normal (SBP<130 and DBP<85 mmHg and not optimal) | 188 | 29 | 3 | 12
  High-normal (SBP<140 DBP<90 mmHg and not normal) | 163 | 92 | 9 | 34
  Stage 1 hypertension (SBP<160 and DBP<100 mmHg | 122 | 73 | 12 | 105
  Stage 2 hypertension (SBP>=160 and DBP>=100 mmHg) | 13 | 8 | 0 | 24

10. Secondary Outcome: Time to First Additional Antihypertensive
Description: Time from first intake of medication to first intake of an antihypertensive other than the study drug
Time Frame: At any point during open-label treatment
Population: Patients from the full analysis set who took additional antihypertensive medication as defined by the investigator. Full analysis set defined as all patients who took at least one dose of study medication and have at least one on treatment BP measurement 20-30 hours post dose
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Total
Number analyzed (Participants) | 218
Days | 85.8 (38.4)

11. Secondary Outcome: Patients Requiring Additional Antihypertensive Therapy to Achieve DBP Control
Description: The number of patients with DBP control (DBP<90 mmHg). Last trough DBP measurement before taking additional antihypertensive compared to last trough DBP taken on treatment
Time Frame: At any point during open-label treatment
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Pre-antihypertensive: Yes (DBP<90 mmHg) | Pre-antihypertensive: No (DBP>=90 mmHg) | Pre-antihypertensive: Total
Number analyzed (Participants) | 12 | 206 | 218
Participants
  Post-antihypertensive: Yes (DBP<90 mmHg) | 10 | 100 | 110
  Post-antihypertensive: No (DBP>=90 mmHg) | 2 | 106 | 108
  Post-antihypertensive: Total | 12 | 206 | 218

12. Secondary Outcome: Additional Reduction in DBP by Use of Additional Antihypertensive Therapy
Description: Difference in trough DBP from last visit before add-on therapy and last visit during 1235.7
Time Frame: At any point during open-label treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Total
Number analyzed (Participants) | 218
mmHg | -5.73 (7.65)

13. Secondary Outcome: Additional Reduction in SBP by Use of Additional Antihypertensive Therapy
Description: Difference in trough SBP from last visit before add-on therapy and last visit during 1235.7
Time Frame: At any point during open-label treatment
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Total
Number analyzed (Participants) | 218
mmHg | -7.53 (11.21)

14. Secondary Outcome: Trough DBP Control Pre- and Post- Uptitration
Description: The number of patients with DBP control (DBP<90 mmHg). Last trough DBP measurement before uptitration to Telmisartan 80mg compared to first trough DBP taken after uptitration
Time Frame: At any point during open-label treatment
Population: Patients from the full analysis set who up-titrated to the higher dose of telmisartan 80 mg and amlodipine 10 mg. Full analysis set defined as all patients who took at least one dose of study medication and have at least one on treatment BP measurement 20-30 hours post dose
Measure: Number; unit: Participants
Arm/Group | Pre-titration: Yes (DBP<90 mmHg) | Pre-titration: No (DBP>=90 mmHg) | Pre-titration: Total
Number analyzed (Participants) | 17 | 361 | 378
Participants
  Post-titration: Yes (DBP<90 mmHg) | 17 | 190 | 207
  Post-titration: No (DBP>=90 mmHg) | 0 | 171 | 171
  Post-titration: Total | 17 | 361 | 378

ADVERSE EVENTS:
Time Frame: From day of first dose until one day after last dose
Description: Safety analysis treatment groups were based upon actual treatment received at the time of the event regardless of add-on antihypertensive. All patients started the study on Telmisartan 40mg and amlodipine 5mg and were up-titrated according to DBP response. Explaining the large number of patients exposed to T40/A5 compared to T80/A5
Arm/Group | Telmisartan 40mg and Amlodipine 5mg | Telmisartan 80mg and Amlodipine 5mg
Serious Adverse Events (participants affected / at risk) | 22/976 | 6/397
Other Adverse Events (participants affected / at risk) | 57/976 | 45/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40mg and Amlodipine 5mg (N=976) | Telmisartan 80mg and Amlodipine 5mg (N=397)
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cronary artery disease (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Cystic lymphangioma (Congenital, familial and genetic disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 1
Typhoid fever (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Hypotonia (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Perpheral artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40mg and Amlodipine 5mg (N=976) | Telmisartan 80mg and Amlodipine 5mg (N=397)
Oedema peripheral (General disorders) | 32 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.